CLINICAL TRIAL: NCT01085968
Title: PC-based Rehabilitation of Motor Planning Deficits in Parkinson Disease
Brief Title: Cognitive Rehabilitation in Parkinson's Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: E7185-R
Record Dates: First submitted 2010-03-10; First posted 2010-03-12 (Estimated); Results first posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Cognitive deficits; fMRI; neuro rehabilitation; Age Matched Controls
MeSH Terms: conditions — Parkinson Disease; Cognition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PD Subjects (Experimental): PD subjects who undergo to PC-based neurorehabilitation intervention. This intervention will train research subjects to improve movement initiation in response to visual stimuli.
  Interventions: Behavioral: PC based training
- Control Subjects (Active Comparator): Age matched controls who undergo to PC-based neurorehabilitation intervention. This intervention will train research subjects to improve movement initiation in response to visual stimuli.
  Interventions: Behavioral: PC based training

INTERVENTIONS:
Behavioral: PC based training — Subjects sit at a computer and type a string of numbers that appears on the screen. As performance improves (# correct), the strings of numbers get longer. They are then instructed to repeat the string from memory. Performing these key entries from memory is a test of internally generated movement initiation.
  Other Names: training

SUMMARY:
We are testing a computer game-style rehabilitation program for people with Parkinson's disease (PD). People with PD often have difficulty with motor planning, such as initiating or starting movements. We believe that our program will improve performance on a movement initiation task as well as on activities of daily living, such as walking, preparing a meal or opening a medicine bottle. We will measure brain function using functional MRI before and after training to identify brain areas that are involved in improved performance. If effective, computer based training will be an inexpensive treatment for motor planning deficits in PD that is free from side effects and easy to administer to a large number of patients.

DETAILED DESCRIPTION:
Our approach is to use PD-based adaptive training to improve performance on IG movement initiation in patients with PD. We have three aims, 1) to systematically evaluate cognitive rehabilitation in people with Parkinson's disease (PD), 2) to examine the neural mechanisms subserving cognitive rehabilitation in PD and 3) to assess the ecological validity of cognitive rehabilitation in PD. We will focus on a single aspect of cognitive function, the decision to initiate a movement. Movements can be internally generated (IG) or externally cued, and motor deficits in PD are typically linked to IG movements. The protocol is designed to drive beneficial neuroplastic changes using a paradigm similar to those that have shown promising results in traumatic brain injury patients. In addition, we will use fMRI to measure activity in underlying basal ganglia-thalamocortical circuits. Finally, because the goal of any research regarding the pathophysiology of disease is to improve the lives of patients with the disease, behavioral and neuropsychological measures will be correlated with fMRI measured functional abnormalities before and after training. Improvement in the initiation of movement has the potential to dramatically improve daily functioning including reducing falls, improving language production and improving proficiency of activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PD dominant on the right side with a Hx of response to dopamine replacement.

Exclusion Criteria:

* Contraindication to MRI
* History of stroke or significant head trauma
* Significant vision impairment
* Hx of brain surgery or claustrophobia
* Medication change <4 weeks
* Atypical PD
* Severe tremor
* Presence of motor fluctuations or dyskinesia
* Significantly impaired limb or joint function
* Significant memory impairment
* Depression or daytime sleepiness

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Disbrow, PhD, Principal Investigator — Overton Brooks VA Medical Center, Shreveport, LA

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be available upon request.

REFERENCES:
- [Result] Disbrow EA, Russo KA, Higginson CI, Yund EW, Ventura MI, Zhang L, Malhado-Chang N, Woods DL, Sigvardt KA. Efficacy of tailored computer-based neurorehabilitation for improvement of movement initiation in Parkinson's disease. Brain Res. 2012 May 3;1452:151-64. doi: 10.1016/j.brainres.2012.02.073. Epub 2012 Mar 9. PMID 22459048

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were assigned to group depending on disease status
Groups:
- PD Subjects: PD subjects
  PC based training: Subjects sit at a computer and type a string of numbers that appears on the screen. They are then instructed to repeat the string from memory. As performance improves (# correct), the strings of numbers get longer.
- Control Subjects: Age matched controls
  PC based training: Subjects sit at a computer and type a string of numbers that appears on the screen. They are then instructed to repeat the string from memory. As performance improves (# correct), the strings of numbers get longer.
Period: Overall Study
Arm/Group | PD Subjects | Control Subjects
Started | 29 | 25
Completed | 19 | 21
Not Completed | 10 | 4

BASELINE CHARACTERISTICS:
Population: Multivariate Analysis of Variance was performed to identify differences across groups in baseline characteristics
Groups:
- Total: Total of all reporting groups
Arm/Group | PD Subjects | Control Subjects | Total
Number analyzed (Participants) | 29 | 25 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.965 (6.450) | 65.56 (6.777) | 66.852 (6.651)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 19 | 15 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 28 | 23 | 51
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 25 | 54

OUTCOME MEASURES:

1. Primary Outcome: Reaction Time and Variability for Movement Task
Description: Before and after computer training outcome measures: left, right, bimanual external cue reaction time; left, right, bimanual external cue error; left, right, bimanual internally generated reaction time; left, right, bimanual internally generated error for four-digit trials.
Time Frame: time of enrollment and 2 months following enrollment (before and after training)
Population: PD Subjects: total number of subjects: 29, 8 withdrew from study, 2 had incomplete data. CO Subjects: total number of subjects: 25, 4 withdrew from study
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | PD Subjects | Control Subjects
Number analyzed (Participants) | 19 | 21
milliseconds
  Before-Left External Cue Reaction Time | 1013.858333 (177.4262864) | 994.94875 (176.9697627)
  Before-Right External Cue Reaction Time | 979.2450877 (199.6872689) | 910.9120833 (170.180081)
  Before-Bimanual External Cue Reaction Time | 1071.54693 (163.2915835) | 1069.631 (168.0096474)
  Before-Left Internally Generated Reaction Time | 763.6505789 (302.5488871) | 708.4873763 (232.2714027)
  Before-Right Internally Generated Reaction Time | 777.4738004 (337.0400281) | 663.6865168 (204.432536)
  Before-Bimanual Internally Generated Reaction Time | 945.8269072 (403.384961) | 774.904215 (206.3438777)
  After-Left External Cue Reaction Time | 723.402193 (197.3197509) | 665.95125 (93.82810385)
  After-Right External Cue Reaction Time | 684.8451754 (187.8980546) | 609.0429167 (93.12353905)
  After-Bimanual External Cue Reaction Time | 730.595614 (209.7713843) | 626.12875 (98.01583054)
  After-Left Internally Generated Reaction Time | 531.5406167 (226.8508076) | 407.7467803 (78.537003)
  After-Right Internally Generated Reaction Time | 532.3444019 (195.9000996) | 402.6036742 (83.0771526)
  After-Bimanual Internally Generated Reaction Time | 575.3801872 (247.1520766) | 432.5232121 (92.77491618)

2. Secondary Outcome: Neuropsychological Measures of Cognitive Function, Including Reaction Time and Time to Completion
Description: Modified Emory Functional Ambulatory Profile (mEFAP); mobility test Task 1: 5 meter walk on hard surface; timed. Task 2: 5 meter walk on carpeted surface, timed. Task 3: Timed up and go; rise from chair, walk 3 meters, walk back, sit down in chair, timed.
  Task 4: Obstacle course, similar to the Timed up and go, with 2 obstacles to be stepped over while walking forward and coming back; timed.
  Task 5: Ascend and descend 5 steps of stairs; timed.
Time Frame: time of enrollment and 2 months following enrollment (before and after training)
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | PD Subjects | Control Subjects
Number analyzed (Participants) | 19 | 21
Seconds
  Before-mEFAP Task 1 | 6.251 (5.849) | 4.897 (0.838)
  Before-mEFAP Task 2 | 6.275 (4.183) | 4.933 (0.792)
  Before-mEFAP Task 3 | 18.853 (15.128) | 14.123 (2.776)
  Before-mEFAP Task 4 | 23.957 (23.470) | 16.320 (3.969)
  Before-mEFAP Task 5 | 9.727 (3.274) | 9.654 (3.974)
  After-mEFAP Task 1 | 6.532 (5.307) | 5.919 (4.015)
  After-mEFAP Task 2 | 6.529 (4.658) | 6.029 (3.927)
  After-mEFAP Task 3 | 20.218 (16.079) | 17.151 (11.656)
  After-mEFAP Task 4 | 22.426 (18.451) | 19.008 (14.091)
  After-mEFAP Task 5 | 10.399 (6.127) | 11.057 (10.976)
  Before-mEFAP Total | 65.034 (49.781) | 49.936 (10.858)
  After-mEFAP Total | 66.105 (49.934) | 59.115 (44.468)

3. Secondary Outcome: Task Errors and Variability
Description: Left, right and bimanual errors in external cue and internally generated tasks for four-digit trials
Time Frame: time of enrollment and 2 months following enrollment (before and after training)
Measure: Mean (Standard Deviation); unit: Number of Errors
Arm/Group | PD Subjects | Control Subjects
Number analyzed (Participants) | 19 | 21
Number of Errors
  Before-Left External Cue Errors | 14.36842105 (26.38014937) | 6.9 (8.540306909)
  Before-Right External Cue Errors | 10 (15.89199659) | 3.85 (4.771350907)
  Before-Bimanual External Cue Errors | 27.21052632 (48.54159608) | 11.3 (12.85997463)
  Before-Left Internally Generated Errors | 3.105263158 (3.016523695) | 1.85 (1.348488433)
  Before-Right Internally Generated Errors | 3.052631579 (3.099707589) | 1.6 (1.602629418)
  Before-Bimanual Internally Generated Errors | 3.578947368 (3.254326854) | 1.65 (1.496487115)
  After-Left External Cue Errors | 4.526315789 (9.026925286) | 0.35 (0.670820393)
  After-Right External Cue Errors | 4.526315789 (9.697470581) | 0.15 (0.670820393)
  After-Bimanual External Cue Errors | 7.421052632 (14.24903813) | 0.6 (1.187655807)
  After-Left Internally Generated Errors | 1.578947368 (2.292882453) | 0.25 (0.444261658)
  After-Right Internally Generated Errors | 1.684210526 (2.906938664) | 0.1 (0.307793506)
  After-Bimanual Internally Generated Errors | 2 (2.666666667) | 0.35 (0.74515982)

4. Secondary Outcome: Functional Dexterity Test (FDT)
Description: Functional Dexterity test (FDT): a motor dexterity measurement for hands. Task: Pick up and flip wooden pegs on a 4x4 pegboard in a zig-zag pattern; timed. Task is performed 2 times per hand Modified Task: Interchange 2 columns of of pegs (4 pegs each side) simultaneously. No flipping is required.
  5 second penalty to time score for 1.) using the pegboard to help with flipping and 2.) supinating of the hand; per occurrence. 10 second penalty to time score for dropping a peg, per occurrence.
Time Frame: time of enrollment and 2 months following enrollment (before and after training)
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | PD Subjects | Control Subjects
Number analyzed (Participants) | 19 | 21
Seconds
  Before-Dominant Hand 1 | 55.048 (37.158) | 41.440 (13.477)
  Before-Dominant Hand 2 | 47.023 (29.848) | 37.627 (18.291)
  Before-Non-dominant Hand 1 | 54.234 (24.115) | 40.585 (18.051)
  Before-Non-dominant Hand 2 | 45.738 (22.573) | 32.193 (11.012)
  Before-Modified Task 1 | 10.034 (2.169) | 10.259 (4.984)
  Before-Modified Task 2 | 9.677 (3.091) | 10.005 (6.149)
  Before-Combined Modified Task | 19.711 (4.324) | 20.263 (8.854)
  Before-Dominant Hand Average | 51.032 (32.445) | 39.533 (12.963)
  Before-Non-dominant Average | 49.987 (19.890) | 36.389 (13.175)
  After-Dominant Hand 1 | 44.831 (25.128) | 35.219 (11.564)
  After-Dominant Hand 2 | 41.261 (28.016) | 29.515 (9.231)
  After-Non-dominant Hand 1 | 46.676 (26.151) | 35.914 (15.678)
  After-Non-dominant Hand 2 | 38.403 (20.954) | 34.533 (14.462)
  After-Modified Task 1 | 9.827 (2.169) | 9.976 (4.811)
  After-Modified Task 2 | 9.508 (4.302) | 7.515 (1.718)
  After-Combined Modified Task | 19.335 (5.969) | 17.492 (5.930)
  After-Dominant Average | 43.046 (25.748) | 32.367 (9.306)
  After-Non-dominant Average | 42.539 (22.706) | 35.224 (14.562)

5. Secondary Outcome: Symbol Digit Modality Test (SDMT)
Description: Symbol Digit Modality Test (SDMT): Participants are given a key of numbers (1-9) corresponding to symbols for reference.
  Task: Participants are given a page of symbols and are instructed to say aloud the number corresponding to each symbol on the page.
  This task is timed for completion and the score is reported as the number of symbol to number matching correct in 90 seconds.
Time Frame: time of enrollment and 2 months following enrollment (before and after training)
Measure: Mean (Standard Deviation); unit: Number of Correct Matches in 90 seconds
Arm/Group | PD Subjects | Control Subjects
Number analyzed (Participants) | 19 | 21
Number of Correct Matches in 90 seconds
  Before-SDMT Number Correct in 90 Seconds | 46.842 (11.644) | 49.286 (8.468)
  After-SDMT Number Correct in 90 Seconds | 48.211 (11.424) | 51.000 (9.338)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for each research participant over the 10-12 week period during which data was collected.
Description: The most likely time that adverse events would be reported was during the 6 weeks of neurorehabilitation training.
Arm/Group | PD Subjects | Control Subjects
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/25
Other Adverse Events (participants affected / at risk) | 0/29 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes